CLINICAL TRIAL: NCT03874351
Title: A Randomized Sham-Controlled Study of Home-Delivered Non-Invasive Neurostimulation for Migraine
Brief Title: A Study of Home-Delivered Neurostimulation for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MJHS Institute for Innovation in Palliative Care (Other)
Collaborators: New York Headache Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19008-01
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Migraine Disorders
Keywords: Migraine;; transcranial direct current stimulation (tDCS); tDCS-Telehealth intervention
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): Twenty minutes of direct current at intensity of 1.5 milliamperes (mA).
  Interventions: Device: non-invasive transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Thirty seconds of direct current at 1.5 mA, followed by 0 mA for the remaining time of the 20-minute stimulation period.
  Interventions: Device: non-invasive transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: non-invasive transcranial direct current stimulation (tDCS) — Active tDCS: transcranial direct current stimulation at intensity 1.5mA for 20 minutes per day on 60 consecutive days, over the area of the dorsolateral prefrontal cortex, using sponge saline-premoisturized electrodes of size 5x5cm, the anode on the left, the cathode on the right.
  Sham tDCS: transcranial direct current stimulation at intensity 1.5mA for 30seconds followed by 0 mA current for remaining time of the 20-minute intervention per day on 60 consecutive days, over the area of the dorsolateral prefrontal cortex, using sponge saline-premoisturized electrodes of size 5x5cm, the anode on the left, the cathode on the right.

SUMMARY:
There is a need for better preventive and abortive therapies for migraine. Previous research has indicated that non-invasive neurostimulation may have prophylactic effects on migraine and improve symptoms and functional outcomes in migraineurs. One such method is a non-invasive transcranial direct current stimulation (tDCS). This double-blind randomized sham-controlled two-parallel-arm study aims to evaluate efficacy and safety of tDCS self-delivered in daily 20-minute applications for 2 months (60 days) by adult migraine patients at home for migraine prevention and migraine symptom management, as compared to sham tDCS application; and to evaluate patients' satisfaction with the procedure.

DETAILED DESCRIPTION:
This study will employ a double-blind randomized sham-controlled two-parallel-arm design and involve 60 adults with migraine. For each participant, the study will involve 3 study visits and last about 90 days (30 days of the baseline followed by 60 days of the tDCS/sham study intervention). A post-study safety monitoring will continue bi-weekly by phone for 30 days after the last tDCS/sham application.

At Visit 1, patients will provide written informed consent and undergo screening for the eligibility. This will be followed by 30 days of baseline at home during which patients will keep daily records (Daily Diaries) of migraine occurrence and provide answers to a set of symptom-related questionnaires. Patients with 4 or more migraine days per month who fully meet the study eligibility criteria at the end of the baseline period will be randomized in double-blind manner into two groups: Group 1 will be randomized to receive active tDCS in daily 20-minute applications for 60 days; Group 2 will be randomized to receive sham tDCS in daily 20-minute applications for 60 days, self-applied at home. Following randomization, patients will continue keeping the Daily Diaries and Visit #2 will be held either in the patient's home or in the research facility, based on the patient's preference. tDCS device will be deployed to the patient and instructions on tDCS use will be provided. The first tDCS/sham self-application by the patient will be done at Visit 2. Daily tDCS/sham self-application by the patient at home and records in the form of Daily Diaries will continue for the rest of the 60-day period. Study staff will be in regular remote contact with the patient via phone and/or HIPAA-compliant videoconferencing. Upon conclusion of the intervention, Visit 3 will be held either in the patient's home or in the research facility, based on the patient's preference. tDCS device will be collected from the patient. Safety monitoring will continue bi-weekly by phone for 30 days after the last tDCS/sham application.

Outcome assessment will be carried out at the end of the baseline, and at Day 30 (the secondary time-point) and Day 60 (the primary time-point) of the tDCS/sham intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years;
* Has episodic or chronic migraine with or without aura, diagnosed according to the International Classification of Headache Disorders 3rd edition (ICHD-3) criteria, for at least the past 12 months;
* Migraine occurring on 4 or more days per month, as documented through the 30-day baseline;
* No change in prophylactic therapy in 3 months preceding the baseline;
* If on antidepressant, blood pressure or epilepsy medication for reason other than migraine, the medication regimen is stable for at least 3 months preceding the baseline; Able to follow instructions in English;
* Understand the informed consent process and provide consent to participate in the study.

Exclusion Criteria:

* History of severe head trauma, brain surgery, implants in the head or neck; history of seizures;
* Skin disorder or skin defects which compromise the integrity or sensitivity of the skin at or near locations where tDCS will be applied;
* Not able to prepare and operate the tDCS device after being instructed in tDCS use;
* Not able to respond to questionnaires and rating scales;
* Concurrent use of another neurostimulation device (such as spinal cord stimulator cardiostimulator, deep brain stimulator, vagus nerve, transcranial magnetic, or supraorbital transcutaneous electric nerve stimulators);
* Concurrent use of Botox or calcitonin gene-related peptide (CGRP) monoclonal antibodies treatments;
* Unstable acute medical condition;
* Any serious, malignant or non-malignant, acute or chronic medical condition or active psychiatric illness that, in the Investigator's opinion, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study;
* Used any investigational drug, biologic, or device within 30 days prior to screening, or 5 half-lives, whichever is longer;
* Taking opioid analgesics or barbiturates on more than 2 days a week;
* Taking medications acting as antagonist on the N-methyl-D-aspartate (NMDA) receptor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Knotkova, PhD, Principal Investigator — MJHS Institute for Innovation in Palliative Care (MJHSPalliative)
Locations (2):
- United States (2):
  - MJHS Institute for Innovation in Palliative Care, New York, New York
  - New York Headache Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the New York Headache Center, New York City, NY, USA, between 3/12/2019 and 3/5/2020.
Pre-assignment Details: Thirty six patients have been identified. Six declined to participate, 14 did not meet the Inclusion/Exclusion criteria. Twenty two proceeded with the study, were randomized and received the study intervention. The first of the twenty-two patients entered the study on 4/22/19; the last patient out completed the study intervention on 4/10/2020, with the last study visit on 4/13/2020 and the last phone follow-up on 5/12/2020.
Groups:
- Active tDCS: The active tDCS will involve 20-minutes of direct current at intensity of 1.5 milliamperes (mA).
  non-invasive transcranial direct current stimulation (tDCS): Non-invasive remotely supervised transcranial direct current stimulation at intensity 1.5mA or sham applied by participants at home for 20 minutes per day on 60 consecutive days, over the area of the dorsolateral prefrontal cortex, using sponge saline-premoisturized electrodes of size 5x5cm, the anode on the left, the cathode on the right.
- Sham tDCS: Sham will include 30 seconds of stimulation at 1.5 mA, followed by 0 mA for the remaining time.
  non-invasive transcranial direct current stimulation (tDCS): Non-invasive remotely supervised transcranial direct current stimulation at intensity 1.5mA or sham applied by participants at home for 20 minutes per day on 60 consecutive days, over the area of the dorsolateral prefrontal cortex, using sponge saline-premoisturized electrodes of size 5x5cm, the anode on the left, the cathode on the right.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 11 | 11
Completed | 7 | 9
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 10 | 5 | 15
  African American | 0 | 2 | 2
  Hispanic | 1 | 2 | 3
  Asian | 0 | 2 | 2
Migraine days per month [Median (Inter-Quartile Range); unit: migraine days per month] — Number of migraine days per month, as reported by participants.
  migraine days per month | 25 [19 to 29] | 17 [9 to 27] | 23 [11 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Migraine Days Per Month
Description: A migraine day is defined as any calendar day on which the patient had onset, continuation, or recurrence of a migraine as recorded in the diary. A migraine is defined as a migraine (with or without aura) lasting at least 30 minutes. Any calendar day on which acute migraine medication is used is counted as a migraine day.
Time Frame: Baseline, Day 30 of the intervention (secondary time point), Day 60 of the intervention (primary time point);
Population: Participants who met the Inclusion/Exclusion criteria for the study.
Measure: Median (Inter-Quartile Range); unit: migraine days per month
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
migraine days per month
  Migraine days per month at day 60 of the intervention (primary outcome) (primary) | -8 [-9 to 0] | -4 [-6 to 0]
  Migraine days per month at day 30 of the intervention (secondary outcome) | -3 [-6 to -1] | -3 [-5 to 0]

2. Secondary Outcome: Percentage of Responders
Description: determined as a percentage of patients having at least 50% reduction of monthly migraine days between the one-month baseline and post-intervention, in each of the two study groups
Time Frame: Day 60 of the intervention
Population: Participants who met the Inclusion/Exclusion criteria of the study
Measure: Number; unit: percentage of participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
percentage of participants | 18.18 | 36.36

3. Secondary Outcome: Migraine Attack Frequency
Description: Median change in number of attacks per 30-day period, determined from the patients' diaries
Time Frame: Baseline, Day 30 of the intervention, Day 60 of the intervention
Population: Participants who met the Inclusion/Exclusion criteria of the study.
Measure: Median (Inter-Quartile Range); unit: migraine attacks per month
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
migraine attacks per month
  Migraine attack frequency at day 60 of the interrvention | -1 [-3 to 0] | -2 [-4 to -1]
  Migraine attack frequency at day 30 of the intervention | 1 [0 to 2] | 0 [-1 to 0]

4. Secondary Outcome: Acute Medication Use
Description: Acute antimigraine drug use per month determined from the patient's diaries. Median change in number of days on which an acute medication was used.
Time Frame: Baseline, Day 30 of the intervention, Day 60 of the intervention
Population: Participants who met the Inclusion/Exclusion criteria of the study
Measure: Median (Inter-Quartile Range); unit: Days/month
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
Days/month
  Acute antimigraine drug use - day 30 of the intervention | -1 [-3 to 0] | -1 [-4 to 0]
  Acute antimigraine drug use - day 60 of the intervention | -2 [-4 to 0] | -2 [-9 to 0]

5. Secondary Outcome: Change in Headache Attack Intensity Median Change in NRS From Headache Days in a 30 Day Period
Description: Determined from the 11-point [0-10] Pain Numerical Rating Scale (Pain NRS) on migraine days in the patients' diaries. Higher ratings on the Pain NRS reflect higher intensity of pain.
Time Frame: Baseline, Day 30 of the intervention, Day 60 of the intervention;
Population: Participants who met the Inclusion/Exclusion criteria of the study.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
Score on a scale
  Change in headache attack intensity - day 30 of the intervention | 0 [0 to 0] | -1 [-1 to 0]
  Change in headache attack intensity - day 60 of the intervention | -1 [-2 to 0] | -1 [-1 to 0]

6. Secondary Outcome: Change in Quality of Life: The Migraine Specific Quality of Life Questionnaire (MSQ)
Description: Determined from ratings on the migraine-specific MSQ questionnaire. The questionnaire consists of 14 items, each rated on a scale 1-6, with the total score ranging between 14 and 84. Higher scores reflect poorer quality of life.
Time Frame: Baseline, Day 30 of the intervention, Day 60 of the intervention;
Population: Participants who met the Inclusion/Exclusion criteria of the study.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
Score on a scale
  Change in quality of life - day 30 of the intervention | -11 [-18 to -5] | -7 [-11 to -2]
  Change in quality of life - day 60 of the intervention | -12 [-18 to -10] | -8 [-25 to -1]

7. Secondary Outcome: Change in Depressive Symptoms
Description: Determined from the Hamilton Depression Scale (HamD) that consists of 21 items with numerically rated responses ranging 0-2 or 0-4. Higher Ham-D score reflects more severe depression.
Time Frame: Baseline, Day 30 of the intervention, Day 60 of the intervention;
Population: Participants who met the Inclusion/Exclusion criteria of the study
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
Score on a scale
  Change in depressive symptoms - day 30 of the intervention | -4 [-7 to -3] | -2 [-4 to 0]
  Change in depressive symptoms - day 60 of the intervention | -5 [-7 to -4] | -3 [-6 to 0]

8. Secondary Outcome: Tolerability of the Study Intervention: Number of Side Effects and Adverse Events
Description: Determined as number of side effects and adverse events related, probably related or possibly related to the study intevention
Time Frame: from Day 1 of the study intervention to the end of the safety follow-up thirty days after the last tDCS application
Population: Participants who met the Inclusion/Exclusion criteria of the study.
Measure: Number; unit: events
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
events | 3 | 0

9. Secondary Outcome: Patient's Satisfaction: 8-item tDCS User Survey
Description: Patient's satisfaction with the study intervention determined from the 8-item tDCS User Survey at the end of the intervention. Each item of the Survey is a brief statement and a respondent indicates if s/he Strongly Agree, Agree, Neither Agree or Disagree, Disagree or Strongly Disagree with the statement. Higher number of Agree/Strongly Agree ratings reflects higher satisfaction with the tDCS procedure.
Time Frame: Day 60 of the intervention
Population: Participants who met the Inclusion/Exclusion criteria of the study
Measure: Number; unit: number of Agree/Strongly Agree ratings
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 11 | 11
number of Agree/Strongly Agree ratings | 41 | 57

ADVERSE EVENTS:
Time Frame: Three months (through the two-month neurostimulation period plus 30 days after the last stimulation).
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS (N=11) | Sham tDCS (N=11)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03874351/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03874351/SAP_002.pdf